CLINICAL TRIAL: NCT01076816
Title: Dexmedetomidine Pharmacokinetics-pharmacodynamics in Mechanically Ventilated Children With Single-organ Respiratory Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor inclusion rate.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/518
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Respiratory Failure
Keywords: Patients with single-organ failure in need of mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Dexmedetomidine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine will be given max 48h. In case analgosedation is still needed after stop of the dexmedetomidine infusion, the treatment is switched to conventional analgosedation regimens.
  Additional drugs are given to every inadequately sedated patient (assessed by regular Comfort scoring). In case of oversedation or adverse drug events (hypotension, bradycardia), a downtitration (or stop) of the dexmedetomidine infusion is needed.
Procedure: Vital signs — systolic and diastolic blood pressure, heart rate, respiratory rate,oxygen saturation, temperature are assessed baseline and at least per hour reassessed after starting the dexmedetomidine.
Procedure: blood sampling — Blood sampling for pharmacokinetic modelling is limited to a maximum of 1,8 ml/kg (in line with the EMEA guidelines on maximum blood sampling in children). Pharmacokinetic parameters and influence of covariates on these parameters will be assessed by a population pharmacokinetic approach.

SUMMARY:
Currently, dexmedetomidine is approved by the United States Food and Drug Administration (FDA) for short-term analgosedation (<24h) in mechanically-ventilated critical care adult patients and sedation of non-intubated adult patients prior to and/or during surgical and other procedures. Trials are underway to investigate its pharmacokinetics, clinical efficacy and safety in long-term use. Clinical experience with dexmedetomidine in the paediatric population is limited. Moreover, during childhood many developmental changes take place with consequences on drug exposure and drug response. Finally, critical illness itself can affect drug pharmacokinetics and -dynamics. Therefore, we cannot simply extrapolate adult data for use in children but we are in need of data on pharmacokinetics and pharmacodynamics in every paediatric subpopulation.

ELIGIBILITY:
Inclusion Criteria:

* patients (m/f) admitted to the paediatric intensive care unit
* expected to require at least 24h of mechanical ventilation
* patient age : 1 month-15 years
* patients with single-organ respiratory failure

Exclusion Criteria:

* patients with neurologic conditions that prohibit an evaluation of adequate analgosedation
* no arterial catheter in place at inclusion
* patients who have received another investigational drug within 30 days
* patients on continuous infusion with neuromuscular blockers
* patients with a life expectancy <72h
* patients with a known allergy to lorazepam, midazolam and/or morphine
* heart block
* pre-existing bradycardia
* hemodynamically unstable patients (Wernovsky index > 16 points) after full fluid replacement with crystalloid
* patients with significant renal insufficiency (creatinine plasma level 1 month-5 year : > 1 mg/dl ; 5-10 years : >1.2 mg/dl; > 10 years : > 1.5 mg/dl)
* patients with significant hepatic insufficiency (aspartate aminase >950 UI/L and prothrombin time < 60 or INR >1.4)
* previous treatment with α2-adrenoreceptor agonist clonidine within 14 days

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of dexmedetomidine infusion in mechanically ventilated children with single-organ respiratory failure | 48 hours
covariates contributing to a variability in exposure and response to dexmedetomidine | 48 hours

SECONDARY OUTCOMES:
preliminary knowledge on the level of sedation provided by dexmedetomidine | 48 hours
preliminary knowledge of safety issues | 48 hours
  systolic and diastolic blood pressure, heart rate, respiratory rate, oxygen saturation, temperature are assessed baseline and at least per hour reassessed after starting the dexmedetomidine infusion
knowledge of the contribution of the CYP2A6 and UDP-glucuronosyltransferase genotype (covariate) to the variability in exposure and response to dexmedetomidine | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pieter De Cock, Pharm.D, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: website of University Hospital Ghent — http://www.uzgent.be